CLINICAL TRIAL: NCT06388928
Title: Effect of Menstrual Cycle on the Manual Dexterity of Female Dentists
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Amira Ibrahim Hassanein Abdel-aal, Assistant lecturer, Faculty of Physical Therapy, Horus University, Cairo University
Other Study IDs: P.T.REC/012/004596
Record Dates: First submitted 2024-01-17; First posted 2024-04-29 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-01

CONDITIONS: Menstrual Cycle; Manual Dexterity
Keywords: Menstrual Cycle; Manual Dexterity; Female Dentists

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- This study was assigned as a single group.: All participants, assigned as one group, were assessed as regards the manual dexterity at three different phases of the menstrual cycle (menstrual phase, ovulation phase, and mid-luteal phase).

SUMMARY:
The aim of this observational study was to investigate the effect of the menstrual cycle on the manual dexterity of female dentists.

This study was conducted to answer the following question:

- Is there any effect of the menstrual cycle on the manual dexterity of female dentists?

ELIGIBILITY:
Inclusion Criteria:

* All participants were nulliparous female dentists having a regular menstrual cycle which was confirmed by using a calendar of three consecutive menstrual cycles.
* Their ages ranged from 25 to 35 years old.
* Their BMI was within the normal range (18.5 to 24.9 kg/m²).

Exclusion Criteria:

* Pregnant female dentists.
* Irregular menstrual cycle and any type of hormonal therapy that may affect normal hormonal level fluctuation.
* History of either orthopedic or neurologic diseases causing functional defects of hand strength such as fracture, carpal tunnel syndrome, or De-Quervain's syndrome.
* Upper limb or hand surgery.
* History of systemic diseases like diabetes mellitus.

Ages: 25 Years to 35 Years | Sex: Female
Age Groups: Adult
Gender Based: Yes
Study Population: Forty-five nulliparous female dentists, with at least one year of practice of the manual work, participated in this study. They were recruited from the outpatient clinic of the Faculty of Dentistry, Horus University, and from private dental clinics.
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2023-07-09 (Actual); Primary Completion 2023-12-26 (Actual); Study Completion 2023-12-26 (Actual)

PRIMARY OUTCOMES:
Manual dexterity assessment | Assessment of the female dentists' manual dexterity was performed from July 2023 to December 2023
  Purdue pegboard test (Lafayette, IN 47093 USA, Model 32020A) was used to measure the participants' unimanual and bimanual hand dexterity.

CONTACTS AND LOCATIONS:
Overall Officials: Amira I Hassanein, Principal Investigator — Cairo University
Locations (1):
- Horus University, Damietta, Egypt

IPD SHARING:
Plan to Share IPD: Undecided